CLINICAL TRIAL: NCT02983227
Title: A Phase II Open-Label Extension Study of Patients Previously Enrolled in Study GA29350 to Evaluate the Long-Term Safety and Efficacy of GDC-0853 in Patients With Moderate to Severe Rheumatoid Arthritis
Brief Title: A Study to Evaluate the Long-Term Safety and Efficacy of GDC-0853 in Participants With Moderate to Severe Rheumatoid Arthritis Enrolled in Study GA29350
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GA30067; 2016-000498-19 (EudraCT Number)
Record Dates: First submitted 2016-11-29; First posted 2016-12-06 (Estimated); Results first posted 2020-08-03 (Actual); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — fenebrutinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GDC-0853 (200mg BID) Cohort 1 (Experimental): Participants received GDC-0853 orally twice daily (BID) for 52 weeks, after completing 12 weeks in Cohort 1 of Study GA29350. Cohort 1 participants in GA29350 were enrolled with moderate to severe active Rheumatoid Arthritis (RA) and an inadequate response to previous methotrexate (MTX) therapy and then randomized to 12 weeks of GDC-0853 (50 mg daily, 150 mg daily, or 200 mg BID), adalimumab, or placebo.
  Interventions: Drug: GDC-0853
- GDC-0853 (200mg BID) Cohort 2 (Experimental): Participants received GDC-0853 orally twice daily (BID) for 52 weeks, after completing 12 weeks in Cohort 2 of Study GA29350. Cohort 2 participants in GA29350 were enrolled with moderate to severe active Rheumatoid Arthritis (RA) and an inadequate response to one or two tumor necrosis factor (TNF) inhibitors and methotrexate (MTX) therapy, and then randomized to 12 weeks of GDC-0853 (200 mg BID) or placebo.
  Interventions: Drug: GDC-0853

INTERVENTIONS:
Drug: GDC-0853 — GDC-0853 was administered orally at a dose of 200mg, as per the dosing schedules described above.
  Other Names: RO7010939

SUMMARY:
A study to evaluate the long-term safety and efficacy of GDC-0853 in participants with moderate to severe active Rheumatoid Arthritis (RA) who have completed 12 weeks of study treatment in Study GA29350. Eligible participants from Study GA29350 who elect to participate will receive treatment with GDC-0853 twice daily (BID) in an open-label fashion for 52 weeks, followed by a safety follow-up period of 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Completion of treatment as specified in Study GA29350, including completion of the Day 84 study visit assessments
* Acceptable safety and tolerability during Study GA29350 as determined by the investigator or Medical Monitor
* Have not received any prohibited medications in Study GA29350
* While taking methotrexate, must be willing to receive oral folic acid (at least 5 milligrams per week [mg/week])
* If receiving oral corticosteroids (less than or equal to [</=] 10 milligrams per day [mg/day] prednisone or equivalent) and/or non-steroidal anti-inflammatory drugs, doses have remained stable for the duration of Study GA29350

Exclusion Criteria:

* Met protocol defined treatment stopping criteria during Study GA29350
* Treatment with any investigational agent (i.e., other than study drug) or live/attenuated vaccine or any other prohibited medication during Study GA29350 or since the last administration of study drug in Study GA29350
* In the opinion of the investigator, any new (since initially enrolling in the Phase II Study GA29350), significant, uncontrolled comorbidity that would increase the risk to the participant in Study GA30067
* Pregnant or lactating, or intending to become pregnant during the study
* Participants who experienced a de novo or reactivated serious viral infection such as hepatitis B virus (HBV), hepatitis C virus (HCV), or human immunodeficiency virus (HIV) during the Phase II Study GA29350
* Any major episode of infection requiring hospitalization or treatment with intravenous antibiotics during the Phase II Study GA29350
* Participants who developed a malignancy during the Phase II Study GA29350
* 12-lead electrocardiogram (ECG) on Day 84 in Study GA29350 that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results
* Current treatment with medications that are well known to prolong the QT interval

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 496 (Actual)
Dates: Start 2016-11-30 (Actual); Primary Completion 2019-07-17 (Actual); Study Completion 2019-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (104):
- United States (11):
  - Arizona Arthritis & Rheumatology Associates, P.C., Glendale, Arizona
  - Medvin Clinical Research, Covina, California
  - TriWest Research Associates, LLC, El Cajon, California
  - Saint Jude Heritage Medical Grp, Fullerton, California
  - RASF-Clinical Research Center, Boca Raton, Florida
  - Clinical Research of West Florida, Clearwater, Florida
  - Medication Management, Greensboro, North Carolina
  - Oregon Health & Science Uni, Portland, Oregon
  - Metroplex Clinical Research Centre, Dallas, Texas
  - Baylor Research Inst., Dallas, Texas
  - Accurate Clinical Research, Houston, Texas
- Argentina (11):
  - Instituto de Investigaciones Clinicas-Mar del Plata, Buenos Aires
  - APRILLUS, Buenos Aires
  - Instituto centenario, Buenos Aires
  - Centro de Investigacion en Enfermedades Reumaticas CIER, Ciudad Autonoma Buenos Aires
  - Expertia S.A- Mautalen Salud e Investigación, Ciudad Autonoma Buenos Aires
  - CCBR - Buenos Aires - AR; AxisMed SRL, Ciudad Autonoma Buenos Aires
  - ILAIM-CEOM Inst. Latinoamericano de Inv. Medicas, Córdoba
  - Centro de Investigaciones Medicas Mar Del Plata, Mar del Plata
  - Instituto de Investigaciones Clinicas, Rosario
  - CER San Juan Centro Polivalente de Asistencia e Investigacion Clinica, San Juan
  - Centro Medico Privado de Reumatologia; Reumathology, San Miguel
- Brazil (7):
  - CIP - Centro Internacional de Pesquisa X; Pesquisa Clinica, Goiânia, Goiás
  - CMiP - Centro Mineiro de Pesquisa*X*, Juiz de Fora, Minas Gerais
  - Centro de Estudos em Terapias Inovadoras - CETI, Curtiba, Paraná
  - CCBR Brasil Centro de Pesquisas e Análises Clínicas Ltda., Rio de Janeiro, Rio de Janeiro
  - LMK Serviços Médicos S/S, Porto Alegre, Rio Grande do Sul
  - CAEP - Centro Avancado de Estudos e Pesquisas Ltda., Campinas, São Paulo
  - IMA Brasil - Instituto de Medicina Avancada, São Paulo, São Paulo
- Bulgaria (9):
  - MHAT "Eurohospital" - Plovdiv, OOD; Internal Department, Plovdiv
  - UMHAT "Kaspela", EOOD, Plovdiv
  - Medizinski Zentrar-1-Sevlievo EOOD, Sevlievo
  - MHAT "Hadzhi Dimitar", OOD, Sliven
  - Medical Center Excelsior OOD, Sofia
  - NMTH "Tsar Boris III", Sofia
  - DCC "Alexandrovska", EOOD; Clinic of Neurology, Sofia
  - MC "Synexus - Sofia", EOOD, Sofia
  - UMHAT "SofiaMed", OOD; Department of Neurology, Sofia
- Colombia (3):
  - Centro de Investigacion Medico Asistencial S.A.S, Barranquilla
  - Centro de Investigacion en Reumatologia y Especialdades Medicas SAS. CIREEM, Bogotá
  - Riesgo de Fractura S.A., Bogotá
- Mexico (9):
  - Consultorio Medico en Fundacion el Hospitalito de morelos A.C., Cuernavaca, Morelos
  - Centro de Investigacion en Reumatologia, Mérida, Yucatán
  - Consultorio Particular del Dr. Miguel Cortes Hernandez, Cuernavaca
  - Centro de Investigacion de Tratam Innovadores de Sin SC, Culiacán
  - Centro de Investigacion en Enfermedades Reumaticas y Osteoporosis, Mexicali
  - Centro de Investigacion Clínica GRAMEL S.C, México
  - Policlinica Medica de Queretaro S.C., Querétaro
  - Clinical Research Institute, Tlalnepantla
  - Unidad de Enfermedades Reumaticas y Cronicodegenerativas, Torreón
- Poland (9):
  - NZOZ ZDROWIE Osteo-Medic, Bialystok
  - Szpital Uniwersytecki; nr 2 im. Dr J. Biziela, Bydgoszcz
  - Centrum Medyczne Pratia Katowice I, Katowice
  - CCBR - Lodz - PL, Lodz
  - ETYKA Osrodek Badan Kliniczynch, Olsztyn
  - Ai Centrum Medyczne Sp. Z O.O Sp.K., Poznan
  - Medycyna Kliniczna, Warsaw
  - Centrum Medyczne AMED, Warsaw
  - KO-MED Centra Kliniczne Zamosc, Zamość
- Russia (19):
  - Federal State Budgetary Scientific Institution Research Institute of Rheumatology V.A. Nasonova, Moscow, Moscow Oblast
  - SBIH of Moscow "City Clinical Hospital # 1 n. a. N. I. Pirogov", Moscow, Moscow Oblast
  - SPb SBIH "Clinical Rheumatological Hospital # 25", Saint Petersburg, Sankt-Peterburg
  - Sanavita LLC, Saint Petersburg, Sankt-Peterburg
  - LLC Medical Sanitary Unit, Saint Petersburg, Sankt-Peterburg
  - Center of Family Medicine LC, Yekaterinburg, Sankt-Peterburg
  - SBHI of Yaroslavl Region Clinical Hospital #3, Yaroslavl, Volgograd Oblast
  - SMMIH "Chelyabinsk Regional Clinical Hospital", Chelyabinsk, Voronez
  - SBIH of Yaroslavl region " Regional Clinical Hospital "; Therapy, Yaroslavl, Yaroslavl Oblast
  - SAHI of Kem. "Regional Clinical Hospital for War Veterans", Kemerovo
  - OOO Family Polyclinic, Korolev, Moscow Region
  - Practical Medicine, Moscow
  - Limited Liability Company "Centre of Medical Common Practice", Novosibirsk
  - Ultramed, Omsk
  - SEIHPE Saratov State Medical University n.a. V.I. Razumovskiy, Saratov
  - NIH "Departmental Hospital on Station Smolensk of OJSC "Russian Railways", Smolensk
  - Siberian State Medical University, Tomsk
  - SHI Ulyanovsk Reg Clinical Hospital, Ulyanovsk
  - Territorial Clinical Hospital #2, Vladivostok
- Serbia (5):
  - Institute of Rheumatology, Belgrade
  - Clinical Center Kragujevac, Kragujevac
  - Institute of Treatment and Rehabilitation "Niska Banja", Niška Banja
  - Special hospital for rheumatic diseases Novi Sad, Novi Sad
  - General Hospital "Dr Laza K. Lazarevic" Sabac, Šabac
- Ukraine (21):
  - MI of Healthcare Kyiv RCH P.L. Shupyk NMA of PGE, Kyiv, Chernihiv Governorate
  - CI of Healthcare Kharkiv CCH #8 Dept of Therapy Kharkiv MA of PGE of MOHU, Kharkiv, Kharkiv Governorate
  - CI of TRC, Ternopil, Kherson Governorate
  - Regional CH Dep of Rheumatology SHEI Ivano-Frankivsk NMU, Ivano-Frankivsk, KIEV Governorate
  - SI NSС M.D. Strazhesko Institute of Cardiology of NAMSU, Kyiv, KIEV Governorate
  - Medical Center of Revmotsentr LLC, Kyiv, KIEV Governorate
  - Medical Center of Limited Liability Company Medical Clinic Blagomed, Kyiv, KIEV Governorate
  - Med Center of International Institute of Clinical Trials LLC; Medical Center "OK!Clinic+", Kyiv, KIEV Governorate
  - Lviv Regional Clinical Hospital Dept of Rehmuaatology D. Halytskyi Lviv NMU, Lviv, KIEV Governorate
  - CH of State Border Service of Ukraine (Military Base 2522); Dept of Therapy, D.Halytskyi Lviv NMU, Lviv, KIEV Governorate
  - A.Novak Transcarpathian Regional Clinical Hospital, Uzhhorod, KIEV Governorate
  - National Pirogov Memorial Medical University, Vinnytsia, Podolia Governorate
  - Railway Transp DCH of HealthCenter Branch of PJSC Ukr Railway Dept of Rheumatology, Dnipro, Tavria Okruha
  - City Clinical Hospital #9 Dept of Therapy SI Zaporizhzhia MA of PGE of MoHU, Zaporizhzhia, Tavria Okruha
  - CI City Hospital #1, Zaporizhzhia, Tavria Okruha
  - CI Lutsk CCH Volyn Regional Center of Cardiovascular Pathology and Thrombolysis, Lutsk, Volhynian Governorate
  - GI L.T.Malaya Therapy National Institute of the NAMS of Ukraine, Kharkiv
  - CNI Consultative and Diagnostic Center of Desnianskyi District of Kyiv, Kyiv
  - M.V. Sklifosovsky Poltava RCH Dept of Rheumatology HSEIU UMSA, Poltava
  - CI City Hospital #7, Zaporizhzhia
  - CI Zaporizhzhia Regional Clinical Hospital of ZRC, Zaporizhzhia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 138 centers in 19 countries.
Pre-assignment Details: 496 participants were enrolled into this OLE study and were included in the ITT and Safety populations.
Period: Overall Study
Arm/Group | GDC-0853 (200mg BID) Cohort 1 | GDC-0853 (200mg BID) Cohort 2
Started | 410 | 86
Completed | 351 | 72
Not Completed | 59 | 14
Not completed — Adverse Event | 21 | 3
Not completed — Death | 3 | 0
Not completed — Lack of Efficacy | 8 | 1
Not completed — Lost to Follow-up | 3 | 0
Not completed — Multiple Reasons | 2 | 1
Not completed — Physician Decision | 3 | 1
Not completed — Withdrawal by Subject | 19 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GDC-0853 (200mg BID) Cohort 1 | GDC-0853 (200mg BID) Cohort 2 | Total
Number analyzed (Participants) | 410 | 86 | 496
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.9 (11.7) | 53.5 (12.5) | 50.5 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 334 | 64 | 398
  Male | 76 | 22 | 98
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino | 136 | 30 | 166
  Not Hispanic or Latino | 267 | 56 | 323
  Not Stated | 2 | 0 | 2
  Unknown | 5 | 0 | 5
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaska native | 27 | 11 | 38
  Asian | 1 | 0 | 1
  Black or African American | 7 | 2 | 9
  Multiple | 7 | 2 | 9
  Unknown | 3 | 0 | 3
  White | 365 | 71 | 436

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events (AEs)
Description: An Adverse Event (AE) was considered any unfavorable and unintended sign, symptom, or disease associated with the use of the study drug, whether or not considered related to the study drug. Preexisting conditions that worsened during the study were reported as adverse events.
Time Frame: Day 1 up until 8 weeks after the last dose of study drug (up to 1 year, 2 months)
Population: The Safety-Evaluable Population was defined as all participants who received any study drug and had at least one assessment of safety.
Measure: Number; unit: Percentage
Arm/Group | GDC-0853 (200mg BID) Cohort 1 | GDC-0853 (200mg BID) Cohort 2
Number analyzed (Participants) | 410 | 86
Percentage | 60.2 | 57.0

2. Primary Outcome: Percentage of Participants Achieving American College of Rheumatology 50% (ACR50) Response at Week 52
Description: ACR50 response is defined as a ≥ 50% improvement (reduction) compared with baseline for both total joint count-68 joints (TJC68) and swollen joint count-66 joints (SJC66), as well as for three of the additional five ACR core set variables: Patient's Assessment of Pain over the previous 24 hours: using a Visual Analog Scale (VAS) left end of the line 0=no pain to right end of the line 100=unbearable pain; Patient's Global Assessment of Disease Activity and Physician's Global Assessment of Disease Activity over the previous 24 hours using a VAS where left end of the line 0=no disease activity to right end of the line 100=maximum disease activity; Health Assessment Questionnaire: 20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities, 0=without difficulty to 3=unable to do; and acute-phase reactant [either C-reactive protein or Erythrocyte Sedimentation Rate].
Time Frame: Week 52
Population: The Intent-To-Treat (ITT) Population was defined as all eligible participants enrolled in this OLE study.
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | GDC-0853 (200mg BID) Cohort 1 | GDC-0853 (200mg BID) Cohort 2
Number analyzed (Participants) | 410 | 86
Percentage | 57.1 [52.28 to 61.86] | 50.0 [39.43 to 60.57]

3. Secondary Outcome: Percentage of Participants Achieving ACR50 Response up to Week 12
Description: as for outcome 2
Time Frame: Weeks 4, 8 and 12
Population: The Intent-To-Treat (ITT) Population was defined as all eligible participants enrolled in this OLE study.
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | GDC-0853 (200mg BID) Cohort 1 | GDC-0853 (200mg BID) Cohort 2
Number analyzed (Participants) | 410 | 86
Percentage
  Week 4 | 37.1 [32.40 to 41.75] | 29.1 [19.47 to 38.67]
  Week 8 | 42.4 [37.65 to 47.22] | 34.9 [24.81 to 44.96]
  Week 12 | 45.6 [40.79 to 50.43] | 39.5 [29.20 to 49.87]

4. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 20% (ACR20) Response
Description: ACR20 response is defined as a ≥ 20% improvement (reduction) compared with baseline for both total joint count-68 joints (TJC68) and swollen joint count-66 joints (SJC66), as well as for three of the additional five ACR core set variables: Patient's Assessment of Pain over the previous 24 hours: using a Visual Analog Scale (VAS) left end of the line 0=no pain to right end of the line 100=unbearable pain; Patient's Global Assessment of Disease Activity and Physician's Global Assessment of Disease Activity over the previous 24 hours using a VAS where left end of the line 0=no disease activity to right end of the line 100=maximum disease activity; Health Assessment Questionnaire: 20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities, 0=without difficulty to 3=unable to do; and acute-phase reactant [either C-reactive protein or Erythrocyte Sedimentation Rate]
Time Frame: Weeks 4, 8, 12, 24, 36 and 52
Population: The Intent-To-Treat (ITT) Population was defined as all eligible participants enrolled in this OLE study.
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | GDC-0853 (200mg BID) Cohort 1 | GDC-0853 (200mg BID) Cohort 2
Number analyzed (Participants) | 410 | 86
Percentage
  Week 4 | 69.0 [64.55 to 73.50] | 58.1 [47.71 to 68.57]
  Week 8 | 72.9 [68.63 to 77.23] | 68.6 [58.80 to 78.41]
  Week 12 | 74.4 [70.17 to 78.62] | 73.3 [63.90 to 82.61]
  Week 24 | 75.4 [71.20 to 79.54] | 72.1 [62.61 to 81.57]
  Week 36 | 75.1 [70.94 to 79.31] | 72.1 [62.61 to 81.57]
  Week 52 | 75.4 [71.20 to 79.54] | 68.6 [58.80 to 78.41]

5. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 70% (ACR70) Response
Description: ACR70 response is defined as a ≥ 70% improvement (reduction) compared with Baseline for both total joint count-68 joints (TJC68) and swollen joint count-66 joints (SJC66), as well as for three of the additional five ACR core set variables: Patient's Assessment of Pain over the previous 24 hours: using a Visual Analog Scale (VAS) left end of the line 0=no pain to right end of the line 100=unbearable pain; Patient's Global Assessment of Disease Activity and Physician's Global Assessment of Disease Activity over the previous 24 hours using a VAS where left end of the line 0=no disease activity to right end of the line 100=maximum disease activity; Health Assessment Questionnaire: 20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities, 0=without difficulty to 3=unable to do; and acute-phase reactant [either C-reactive protein or Erythrocyte Sedimentation Rate].
Time Frame: Weeks 4, 8, 12, 24, 36 and 52
Population: The Intent-To-Treat (ITT) Population was defined as all eligible participants enrolled in this OLE study.
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | GDC-0853 (200mg BID) Cohort 1 | GDC-0853 (200mg BID) Cohort 2
Number analyzed (Participants) | 410 | 86
Percentage
  Week 4 | 19.8 [15.90 to 23.61] | 12.8 [5.73 to 19.85]
  Week 8 | 21.7 [17.72 to 25.70] | 17.4 [9.42 to 25.46]
  Week 12 | 23.9 [19.77 to 28.03] | 19.8 [11.35 to 28.18]
  Week 24 | 30.2 [25.80 to 34.69] | 20.9 [12.33 to 29.53]
  Week 36 | 32.2 [27.67 to 36.72] | 25.6 [16.36 to 34.80]
  Week 52 | 36.3 [31.69 to 41.00] | 27.9 [18.43 to 37.39]

6. Secondary Outcome: Disease Activity Score Based on 28-Joints Count and C-Reactive Protein (3 Variables) (DAS28-3 CRP)
Description: The DAS28 score is a measure of the patient's disease activity calculated using the tender joint count (TJC) [28 joints], swollen joint count (SJC) [28 joints], patient's global assessment of disease activity [visual analog scale: 0=no disease activity to 100=maximum disease activity] and the erythrocyte sedimentation rate (ESR) for a total possible score of 0 to approximately 10. Scores below 2.6 indicate best disease control and scores above 5.1 indicate worse disease control. DAS28 Remission is defined as a DAS28 score < 2.6.
Time Frame: Baseline, Weeks 4, 8, 12, 24, 36 and 52
Population: The Intent-To-Treat (ITT) Population was defined as all eligible participants enrolled in this OLE study. Number of participants for whom data were actually collected is indicated for each time point.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | GDC-0853 (200mg BID) Cohort 1 | GDC-0853 (200mg BID) Cohort 2
Number analyzed (Participants) | 406 | 86
Score on a scale
  Baseline | 5.49 (0.85) | 5.59 (0.90)
  Week 4: number analyzed (Participants) | 398 | 83
  Week 4 | 3.64 (1.11) | 4.09 (1.19)
  Week 8: number analyzed (Participants) | 386 | 84
  Week 8 | 3.48 (1.06) | 3.81 (1.15)
  Week 12: number analyzed (Participants) | 378 | 83
  Week 12 | 3.37 (1.09) | 3.73 (1.11)
  Week 24: number analyzed (Participants) | 372 | 82
  Week 24 | 3.16 (1.05) | 3.55 (1.18)
  Week 36: number analyzed (Participants) | 361 | 79
  Week 36 | 3.05 (1.05) | 3.36 (1.06)
  Week 52: number analyzed (Participants) | 349 | 71
  Week 52 | 2.90 (1.03) | 3.17 (1.28)

7. Secondary Outcome: Disease Activity Score Based on 28-Joints Count and C-Reactive Protein (4 Variables) (DAS28-4 CRP)
Description: as for outcome 6
Time Frame: Baseline, Weeks 4, 8, 12, 24, 36 and 52
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | GDC-0853 (200mg BID) Cohort 1 | GDC-0853 (200mg BID) Cohort 2
Number analyzed (Participants) | 391 | 86
Score on a scale
  Baseline: number analyzed (Participants) | 387 | 86
  Baseline | 5.83 (0.88) | 5.95 (0.94)
  Week 4: number analyzed (Participants) | 391 | 83
  Week 4 | 3.70 (1.19) | 4.22 (1.34)
  Week 8: number analyzed (Participants) | 378 | 84
  Week 8 | 3.53 (1.13) | 3.92 (1.25)
  Week 12: number analyzed (Participants) | 373 | 83
  Week 12 | 3.39 (1.14) | 3.81 (1.21)
  Week 24: number analyzed (Participants) | 369 | 82
  Week 24 | 3.18 (1.13) | 3.64 (1.27)
  Week 36: number analyzed (Participants) | 360 | 79
  Week 36 | 3.06 (1.14) | 3.44 (1.21)
  Week 52: number analyzed (Participants) | 348 | 71
  Week 52 | 2.87 (1.09) | 3.22 (1.40)

8. Secondary Outcome: Disease Activity Score Based on 28-Joints Count and Erythrocyte Sedimentation Rate (3 Variables) (DAS28-3 ESR)
Description: as for outcome 6
Time Frame: Baseline, Weeks 4, 8, 12, 24, 36 and 52
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GDC-0853 (200mg BID) Cohort 1 | GDC-0853 (200mg BID) Cohort 2
Number analyzed (Participants) | 404 | 86
Score on a Scale
  Baseline | 6.17 (0.79) | 6.38 (0.88)
  Week 4: number analyzed (Participants) | 397 | 85
  Week 4 | 4.25 (1.16) | 4.80 (1.26)
  Week 8: number analyzed (Participants) | 389 | 83
  Week 8 | 4.04 (1.14) | 4.51 (1.17)
  Week 12: number analyzed (Participants) | 381 | 83
  Week 12 | 3.89 (1.16) | 4.40 (1.11)
  Week 24: number analyzed (Participants) | 375 | 83
  Week 24 | 3.65 (1.08) | 4.15 (1.27)
  Week 36: number analyzed (Participants) | 361 | 79
  Week 36 | 3.46 (1.15) | 3.96 (1.15)
  Week 52: number analyzed (Participants) | 347 | 72
  Week 52 | 3.35 (1.14) | 3.74 (1.31)

9. Secondary Outcome: Disease Activity Score Based on 28-Joints Count and Erythrocyte Sedimentation Rate (4 Variables) (DAS28-4 ESR)
Description: as for outcome 6
Time Frame: Baseline, Weeks 4, 8, 12, 24, 36 and 52
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GDC-0853 (200mg BID) Cohort 1 | GDC-0853 (200mg BID) Cohort 2
Number analyzed (Participants) | 390 | 86
Score on a Scale
  Baseline: number analyzed (Participants) | 385 | 86
  Baseline | 6.48 (0.85) | 6.71 (0.96)
  Week 4: number analyzed (Participants) | 390 | 85
  Week 4 | 4.27 (1.25) | 4.89 (1.41)
  Week 8: number analyzed (Participants) | 381 | 83
  Week 8 | 4.04 (1.23) | 4.58 (1.29)
  Week 12: number analyzed (Participants) | 376 | 83
  Week 12 | 3.87 (1.23) | 4.44 (1.25)
  Week 24: number analyzed (Participants) | 373 | 83
  Week 24 | 3.62 (1.16) | 4.20 (1.37)
  Week 36: number analyzed (Participants) | 360 | 79
  Week 36 | 3.43 (1.24) | 3.99 (1.30)
  Week 52: number analyzed (Participants) | 346 | 72
  Week 52 | 3.27 (1.20) | 3.74 (1.42)

10. Secondary Outcome: Percentage of Participants With Remission Based on Disease Activity Score Based on 28-Joints Count (DAS28)
Description: The DAS28 score is a measure of the patient's disease activity calculated using the tender joint count (TJC) [28 joints], swollen joint count (SJC) [28 joints], patient's global assessment of disease activity [visual analog scale: 0=no disease activity to 100=maximum disease activity] and the erythrocyte sedimentation rate (ESR) for a total possible score of 0 to approximately 10. Scores below 2.6 indicate best disease control and scores above 5.1 indicate worse disease control.
Time Frame: Weeks 4, 8, 12, 24, 36 and 52
Population: The Intent-To-Treat (ITT) Population was defined as all eligible participants enrolled in this OLE study.
Measure: Number; unit: Percentage of Participants
Arm/Group | GDC-0853 (200mg BID) Cohort 1 | GDC-0853 (200mg BID) Cohort 2
Number analyzed (Participants) | 410 | 86
Percentage of Participants
  Week 4 | 8.8 | 7.0
  Week 8 | 10.7 | 8.1
  Week 12 | 13.9 | 8.1
  Week 24 | 17.8 | 14.0
  Week 36 | 22.4 | 11.6
  Week 52 | 25.6 | 23.3

11. Secondary Outcome: Percentage of Participants With Low Disease Activity (LDA) Based on DAS28
Description: The DAS28 score is a measure of the patient's disease activity calculated using the tender joint count (TJC) [28 joints], swollen joint count (SJC) [28 joints], patient's global assessment of disease activity [visual analog scale: 0=no disease activity to 100=maximum disease activity] and the erythrocyte sedimentation rate (ESR) for a total possible score of 0 to approximately 10. Scores below 2.6 indicate best disease control and scores above 5.1 indicate worse disease control. LDAS is defined as DAS28 ≤ 3.2
Time Frame: Weeks 4, 8, 12, 24, 36 and 52
Population: The Intent-To-Treat (ITT) Population was defined as all eligible participants enrolled in this OLE study.
Measure: Number; unit: Percentage of Participants
Arm/Group | GDC-0853 (200mg BID) Cohort 1 | GDC-0853 (200mg BID) Cohort 2
Number analyzed (Participants) | 410 | 86
Percentage of Participants
  Week 4 | 20.0 | 12.8
  Week 8 | 21.2 | 17.4
  Week 12 | 26.6 | 12.8
  Week 24 | 33.7 | 27.9
  Week 36 | 38.3 | 29.1
  Week 52 | 42.2 | 29.1

12. Secondary Outcome: Percentage of Participants With ACR/EULAR Remission
Description: Assessed according to the Boolean based definition (tender joint count =<1, swollen joint count =<1, C-reactive Protein (CRP) =<1, and patient global assessment =<1)
Time Frame: Weeks 4, 8, 12, 24, 36 and 52
Population: as for outcome 6
Measure: Number; unit: Percentage of Participants
Arm/Group | GDC-0853 (200mg BID) Cohort 1 | GDC-0853 (200mg BID) Cohort 2
Number analyzed (Participants) | 401 | 86
Percentage of Participants
  Week 4 | 5.0 | 5.8
  Week 8: number analyzed (Participants) | 397 | 85
  Week 8 | 7.8 | 5.9
  Week 12: number analyzed (Participants) | 390 | 83
  Week 12 | 7.4 | 7.2
  Week 24: number analyzed (Participants) | 378 | 83
  Week 24 | 13.0 | 6.0
  Week 36: number analyzed (Participants) | 366 | 79
  Week 36 | 15.6 | 11.4
  Week 52: number analyzed (Participants) | 353 | 75
  Week 52 | 17.8 | 10.7

13. Secondary Outcome: Change From Baseline in Simplified Disease Activity Index (SDAI)
Description: Simplified Disease Activity Index (SDAI) is the numerical sum of five outcome parameters: TJC and SJC (based on a 28-joint assessment), PtGA and PhGA (based on 0-10 cm VAS, where 0 = no disease activity and 10 = worst disease activity), and CRP. SDAI total score ranges from 0 (no disease activity) to 86 (maximal disease activity), where higher scores represents higher disease activity. The SDAI =< 3.3 indicates disease remission, > 3.4 to 11 indicates low disease activity, > 11 to 26 indicates moderate disease activity, and > 26 indicates high disease activity
Time Frame: Weeks 4, 8, 12, 24, 36 and 52
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GDC-0853 (200mg BID) Cohort 1 | GDC-0853 (200mg BID) Cohort 2
Number analyzed (Participants) | 373 | 84
Score on a Scale
  Week 4: number analyzed (Participants) | 373 | 83
  Week 4 | -24.36 (13.58) | -21.00 (13.49)
  Week 8: number analyzed (Participants) | 362 | 84
  Week 8 | -26.17 (13.58) | -24.06 (13.57)
  Week 12: number analyzed (Participants) | 355 | 83
  Week 12 | -27.91 (12.89) | -25.21 (13.37)
  Week 24: number analyzed (Participants) | 352 | 82
  Week 24 | -29.61 (13.14) | -26.45 (14.17)
  Week 36: number analyzed (Participants) | 342 | 79
  Week 36 | -30.47 (13.72) | -28.22 (14.16)
  Week 52: number analyzed (Participants) | 331 | 71
  Week 52 | -31.69 (13.12) | -29.68 (13.77)

14. Secondary Outcome: Change From Baseline in Clinical Disease Activity Index (CDAI)
Description: CDAI was derived as the sum of the following: tender joint count (TJC), swollen joint count (SJC), participant global assessment (PGA) of disease activity, and physician assessment of disease activity. TJC and SJC were taken as the number of tender and swollen joints, respectively, out of 28 assessed joints. PGA and physician assessment of disease activity were scored 0-100 millimeters (mm) and rounded to the nearest centimeter (cm) on a visual analog scale (VAS), where higher scores indicate greater perceived disease activity. The total CDAI score range was 0-76, where higher scores indicate increased disease activity. Change from baseline at a particular time point was calculated among patients with data available at both baseline and the time point of interest. Negative values indicate improvement/reduction in RA disease activity.
Time Frame: Weeks 4, 8, 12, 24, 36 and 52
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GDC-0853 (200mg BID) Cohort 1 | GDC-0853 (200mg BID) Cohort 2
Number analyzed (Participants) | 374 | 86
Score on a Scale
  Week 4 | -23.41 (13.11) | -19.81 (13.15)
  Week 8: number analyzed (Participants) | 366 | 84
  Week 8 | -25.14 (13.06) | -22.48 (12.59)
  Week 12: number analyzed (Participants) | 360 | 83
  Week 12 | -26.82 (12.31) | -23.82 (12.37)
  Week 24: number analyzed (Participants) | 356 | 83
  Week 24 | -28.52 (12.52) | -25.09 (13.18)
  Week 36: number analyzed (Participants) | 343 | 79
  Week 36 | -29.40 (12.99) | -26.66 (12.98)
  Week 52: number analyzed (Participants) | 332 | 72
  Week 52 | -30.61 (12.43) | -27.43 (13.43)

15. Secondary Outcome: Change From Baseline in Tender/Painful Joint Count Based on 68 Joints
Description: Tender Joint Count: a total of 68 joints will be assessed for tenderness. Each joint is assessed for the presence/absence of tenderness. 68 joints are assessed for tenderness and joints are classified as tender/not tender giving a total possible tender joint count score of 0 to 68. A negative change from Baseline indicated improvement.
Time Frame: Weeks 4, 8, 12, 24, 36 and 52
Population: Intent-to-Treat (ITT) All randomized participants who received any part of an infusion of study medication were included in the ITT analysis. Number of participants for whom data were actually collected is indicated for each time point.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GDC-0853 (200mg BID) Cohort 1 | GDC-0853 (200mg BID) Cohort 2
Number analyzed (Participants) | 406 | 86
Score on a Scale
  Week 4: number analyzed (Participants) | 400 | 86
  Week 4 | -15.02 (12.38) | -13.23 (12.27)
  Week 8: number analyzed (Participants) | 404 | 86
  Week 8 | -16.11 (12.45) | -15.19 (12.59)
  Week 12 | -16.55 (12.39) | -15.99 (12.03)
  Week 24 | -17.96 (12.24) | -16.65 (11.35)
  Week 36 | -18.48 (12.77) | -17.51 (11.60)
  Week 52 | -18.70 (12.99) | -17.73 (11.88)

16. Secondary Outcome: Change From Baseline in Swollen Joint Count Based on 66 Joints
Description: Swollen Joint Count: a total of 66 joints will be assessed for swelling. Each joint is assessed for the presence/absence of swelling. 66 joints were assessed for swelling and joints are classified as swollen/not swollen giving a total possible swollen joint count score of 0 to 66. A negative change from Baseline indicated improvement.
Time Frame: Weeks 4, 8, 12, 24, 36 and 52
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GDC-0853 (200mg BID) Cohort 1 | GDC-0853 (200mg BID) Cohort 2
Number analyzed (Participants) | 406 | 86
Score on a Scale
  Week 4: number analyzed (Participants) | 400 | 86
  Week 4 | -10.20 (8.43) | -7.85 (6.71)
  Week 8: number analyzed (Participants) | 404 | 86
  Week 8 | -10.95 (8.48) | -9.12 (6.65)
  Week 12 | -11.40 (8.22) | -9.08 (6.84)
  Week 24 | -11.93 (8.33) | -9.86 (6.61)
  Week 36 | -12.15 (8.57) | -9.98 (6.96)
  Week 52 | -12.17 (8.55) | -9.59 (8.78)

17. Secondary Outcome: Change From Baseline in Patient's Assessment of Arthritis Pain, Using Visual Analog Scale (VAS) Score
Description: Patient's Assessment of Pain over the previous 24 hours: using a Visual Analog Scale (VAS) left end of the line 0=no pain to right end of the line 100=unbearable pain
Time Frame: Weeks 4, 8, 12, 24, 36 and 52
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GDC-0853 (200mg BID) Cohort 1 | GDC-0853 (200mg BID) Cohort 2
Number analyzed (Participants) | 371 | 86
Score on a Scale
  Week 4 | -30.62 (26.60) | -26.34 (25.98)
  Week 8: number analyzed (Participants) | 365 | 84
  Week 8 | -32.57 (26.77) | -27.21 (23.36)
  Week 12: number analyzed (Participants) | 354 | 83
  Week 12 | -35.68 (26.44) | -29.49 (26.70)
  Week 24: number analyzed (Participants) | 356 | 83
  Week 24 | -37.19 (26.85) | -30.30 (26.42)
  Week 36: number analyzed (Participants) | 343 | 79
  Week 36 | -39.50 (27.20) | -33.14 (27.22)
  Week 52: number analyzed (Participants) | 330 | 72
  Week 52 | -42.40 (26.22) | -38.21 (26.37)

18. Secondary Outcome: Change From Baseline in Patient's Global Assessment of Arthritis, Using VAS Score
Description: Participant-assessed arthritis pain was scored on a 100-mm VAS, where the distance from 0 mm represented the participant's self evaluation of arthritis pain (0 mm=none; 100 mm=very severe). Change from baseline at a particular time point was calculated among patients with data available at both baseline and the time point of interest, where negative change indicated a decrease in participant-assessed arthritis pain.
Time Frame: Weeks 4, 8, 12, 24, 36 and 52
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GDC-0853 (200mg BID) Cohort 1 | GDC-0853 (200mg BID) Cohort 2
Number analyzed (Participants) | 375 | 86
Score on a Scale
  Week 4 | -30.21 (27.47) | -26.03 (24.50)
  Week 8: number analyzed (Participants) | 366 | 84
  Week 8 | -32.67 (26.85) | -28.79 (23.07)
  Week 12: number analyzed (Participants) | 360 | 83
  Week 12 | -35.63 (26.19) | -31.16 (25.32)
  Week 24: number analyzed (Participants) | 356 | 83
  Week 24 | -36.94 (27.23) | -31.76 (25.09)
  Week 36: number analyzed (Participants) | 343 | 79
  Week 36 | -39.40 (26.77) | -33.73 (25.82)
  Week 52: number analyzed (Participants) | 332 | 72
  Week 52 | -42.91 (25.90) | -36.58 (24.74)

19. Secondary Outcome: Change From Baseline in Physician's Global Assessment of Arthritis, Using VAS Score
Description: Physician's assessment of participant's disease activity was scored on a 100-mm VAS, where the distance from 0 mm represented the physician's assessment of the participant's disease activity (0 mm=very good; 100 mm=very poor). Change from baseline at a particular time point was calculated among patients with data available at both baseline and the time point of interest, where negative change from baseline indicated an improvement in physician-assessed disease activity.
Time Frame: Weeks 4, 8, 12, 24, 36 and 52
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GDC-0853 (200mg BID) Cohort 1 | GDC-0853 (200mg BID) Cohort 2
Number analyzed (Participants) | 399 | 86
Score on a Scale
  Week 4 | -37.07 (20.75) | -30.65 (24.09)
  Week 8: number analyzed (Participants) | 390 | 84
  Week 8 | -39.29 (20.30) | -35.32 (22.36)
  Week 12: number analyzed (Participants) | 383 | 83
  Week 12 | -42.23 (20.20) | -37.37 (22.14)
  Week 24: number analyzed (Participants) | 376 | 83
  Week 24 | -44.40 (20.94) | -41.11 (23.86)
  Week 36: number analyzed (Participants) | 362 | 79
  Week 36 | -45.52 (20.76) | -43.13 (24.14)
  Week 52: number analyzed (Participants) | 350 | 72
  Week 52 | -48.57 (19.99) | -44.81 (23.85)

20. Secondary Outcome: Change From Baseline in C-Reactive Protein (CRP) Levels
Description: C-reactive protein is a biological marker of inflammation and is measured in milligrams per decilitre (mg/dL)
Time Frame: Weeks 4, 8, 12, 24, 36 and 52
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: (mg/dL)
Arm/Group | GDC-0853 (200mg BID) Cohort 1 | GDC-0853 (200mg BID) Cohort 2
Number analyzed (Participants) | 398 | 84
(mg/dL)
  Week 4: number analyzed (Participants) | 398 | 83
  Week 4 | -0.95 (2.18) | -1.09 (3.10)
  Week 8: number analyzed (Participants) | 386 | 84
  Week 8 | -1.02 (2.41) | -1.58 (2.60)
  Week 12: number analyzed (Participants) | 378 | 83
  Week 12 | -1.03 (2.21) | -1.40 (3.38)
  Week 24: number analyzed (Participants) | 372 | 82
  Week 24 | -1.03 (2.48) | -1.46 (2.99)
  Week 36: number analyzed (Participants) | 361 | 79
  Week 36 | -1.11 (2.44) | -1.56 (3.04)
  Week 52: number analyzed (Participants) | 349 | 71
  Week 52 | -1.12 (2.55) | -1.81 (2.75)

21. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) Score
Description: The Stanford Health Assessment Questionnaire disability index is a patient-reported outcome used to assess difficulty in performing activities of daily living. It consists of 20 questions referring to eight domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip and common daily activities.
  To respond to each question, a four-level response with higher scores showing larger functional limitations, was chosen. Scoring is as follows with respect to performance of participant's everyday activities: 0 (equals)=without difficulties; 1= with some difficulties; 2=with great difficulties; and 3=unable to perform these actions at all. The composite HAQ-DI score is the mean of the eight domain scores and the score ranges from 0 (no functional impairment) to 3 (maximum functional impairment). A negative change from baseline indicates improvement.
Time Frame: Weeks 4, 8, 12, 24, 36 and 52
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GDC-0853 (200mg BID) Cohort 1 | GDC-0853 (200mg BID) Cohort 2
Number analyzed (Participants) | 360 | 81
Score on a Scale
  Week 4 | -0.70 (0.64) | -0.55 (0.56)
  Week 8: number analyzed (Participants) | 358 | 80
  Week 8 | -0.77 (0.65) | -0.59 (0.62)
  Week 12: number analyzed (Participants) | 358 | 78
  Week 12 | -0.80 (0.67) | -0.60 (0.59)
  Week 24: number analyzed (Participants) | 349 | 78
  Week 24 | -0.83 (0.66) | -0.63 (0.58)
  Week 36: number analyzed (Participants) | 338 | 74
  Week 36 | -0.89 (0.63) | -0.62 (0.66)
  Week 52: number analyzed (Participants) | 323 | 70
  Week 52 | -0.98 (0.64) | -0.69 (0.62)

22. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey (SF-36) Version 2.0 (V2) Scores for Physical and Mental Components
Description: The 36-Item Short Form Health Survey (SF-36v2) is a questionnaire used to assess functional health and well-being and consists of eight domains: Physical Functioning, Role-Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role-Emotional and Mental Health.
  The SF-36v2 is summarized into Physical Component Summary (PCS) and Mental Component Summary (MCS) scores. The PCS and MCS scores range from 0 to 100, with 0=worst score (or quality of life) and 100=best score. A positive change from baseline indicates improvement.
Time Frame: Weeks 12, 24 and 52
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Number on a Scale
Arm/Group | GDC-0853 (200mg BID) Cohort 1 | GDC-0853 (200mg BID) Cohort 2
Number analyzed (Participants) | 356 | 83
Number on a Scale
  Week 12 (Physical Component Score change) | 11.35 (9.13) | 8.22 (8.73)
  Week 12 (Mental Component Score change) | 6.52 (12.98) | 4.74 (11.53)
  Week 24 (Physical Component Score change): number analyzed (Participants) | 350 | 80
  Week 24 (Physical Component Score change) | 12.31 (9.12) | 8.28 (8.53)
  Week 24 (Mental Component Score change): number analyzed (Participants) | 350 | 80
  Week 24 (Mental Component Score change) | 6.63 (13.23) | 6.08 (11.76)
  Week 52 (Physical Component Score change): number analyzed (Participants) | 330 | 72
  Week 52 (Physical Component Score change) | 13.89 (9.32) | 10.42 (8.94)
  Week 52 (Mental Component Score change): number analyzed (Participants) | 330 | 72
  Week 52 (Mental Component Score change) | 7.00 (13.81) | 6.77 (11.60)

23. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) Score
Description: The FACIT-Fatigue Scale consists of 13 items designed to measure the degree of fatigue experienced by the patient in the previous 7 days. For each question, there are five possible responses: 0 (not at all), 1 (a little bit), 2 (somewhat), 3 (quite a bit), 4 (very much).
  A total fatigue score is calculated by summing all items, and possible total scores range from 0 (maximum fatigue) to 52 (no fatigue). A positive change from baseline indicates an improvement in the patient's fatigue (less fatigue).
Time Frame: Weeks 12, 24 and 52
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | GDC-0853 (200mg BID) Cohort 1 | GDC-0853 (200mg BID) Cohort 2
Number analyzed (Participants) | 350 | 83
Score on a Scale
  Week 12 | 11.44 (10.36) | 9.28 (8.51)
  Week 24: number analyzed (Participants) | 347 | 80
  Week 24 | 11.74 (10.75) | 10.41 (8.51)
  Week 52: number analyzed (Participants) | 327 | 72
  Week 52 | 12.87 (10.58) | 10.87 (9.25)

24. Secondary Outcome: Area Under the Concentration Time Curve (AUC) of GDC-0853 at Steady State (AUC,ss)
Description: Population PK model estimated AUC of GDC-0853 at steady-state. AUC was measured in Nanograms (ng) per millilitre(mL)*hour (hr).
Time Frame: Pre-dose (0 hour) on Weeks 0 (Day 1), 4, 12, 24, 36, and 52/early termination
Population: The PK-Evaluable population was defined as all participants that received any fenebrutinib/GDC-0853 and had sufficient data to enable estimation of key PK parameters. Participants who received incorrect therapy different from the intended therapy were summarized in the group according to the therapy actually received.
Measure: Mean (Standard Deviation); unit: Ng/mL*(hr)
Arm/Group | GDC-0853 (200mg BID) Cohort 1 | GDC-0853 (200mg BID) Cohort 2
Number analyzed (Participants) | 388 | 81
Ng/mL*(hr) | 13400 (6930) | 15600 (7850)

25. Secondary Outcome: Minimum Plasma Concentration of GDC-0853 at Steady State (Ctrough,ss)
Description: Population PK model estimated minimal plasma concentration (Ctrough) of GDC-0853 at steady-state (ss).
Time Frame: Pre-dose (0 hour) on Weeks 0 (Day 1), 4, 12, 24, 36, and 52/early termination
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | GDC-0853 (200mg BID) Cohort 1 | GDC-0853 (200mg BID) Cohort 2
Number analyzed (Participants) | 388 | 81
ng/mL | 387 (244) | 467 (285)

26. Secondary Outcome: Plasma Decay Half-Life of GDC-0853 at Steady State (t1/2,ss)
Description: Population PK model estimated plasma decay half life of GDC-0853 at steady-state.
Time Frame: Pre-dose (0 hour) on Weeks 0 (Day 1), 4, 12, 24, 36, and 52/early termination
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | GDC-0853 (200mg BID) Cohort 1 | GDC-0853 (200mg BID) Cohort 2
Number analyzed (Participants) | 388 | 81
hr | 7.94 (3.16) | 9.01 (4.9)

27. Secondary Outcome: Apparent Oral Clearance of GDC-0853 at Steady State (CL/F,ss)
Description: Population PK model estimated apparent oral clearance of GDC-0853 at steady-state.
Time Frame: Pre-dose (0 hour) on Weeks 0 (Day 1), 4, 12, 24, 36, and 52/early termination
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | GDC-0853 (200mg BID) Cohort 1 | GDC-0853 (200mg BID) Cohort 2
Number analyzed (Participants) | 388 | 81
L/hr | 39.5 (12.6) | 35.3 (10.3)

ADVERSE EVENTS:
Time Frame: Day 1 up until 8 weeks after the last dose of study drug (up to 1 year, 2 months).
Description: The Safety-evaluable population was defined as all participants who received any study drug and had at least one assessment of safety. AEs that were entered into the database at the time of the database lock were included in the AE analysis.
Arm/Group | GDC-0853 (200mg BID) Cohort 1 | GDC-0853 (200mg BID) Cohort 2
All-Cause Mortality (participants affected / at risk) | 3/410 | 0/86
Serious Adverse Events (participants affected / at risk) | 26/410 | 4/86
Other Adverse Events (participants affected / at risk) | 22/410 | 4/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GDC-0853 (200mg BID) Cohort 1 (N=410) | GDC-0853 (200mg BID) Cohort 2 (N=86)
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 1 (1)
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 1 (1) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 1 (1) | 0 (0)
ENTEROCOLITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
INFLAMMATORY BOWEL DISEASE (Gastrointestinal disorders) | 1 (1) | 0 (0)
INGUINAL HERNIA (Gastrointestinal disorders) | 1 (1) | 0 (0)
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 1 (1) | 0 (0)
CELLULITIS (Infections and infestations) | 1 (1) | 0 (0)
INFECTION (Infections and infestations) | 1 (1) | 0 (0)
NECROTISING SOFT TISSUE INFECTION (Infections and infestations) | 1 (1) | 0 (0)
OSTEOMYELITIS (Infections and infestations) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1)
PYELONEPHRITIS (Infections and infestations) | 1 (1) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0)
HEAD INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
HIP FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
MULTIPLE INJURIES (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
HEPATIC ENZYME INCREASED (Investigations) | 1 (1) | 0 (0)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
LUNG CARCINOMA CELL TYPE UNSPECIFIED STAGE IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
ISCHAEMIC STROKE (Nervous system disorders) | 1 (1) | 0 (0)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 1 (1) | 0 (0)
VERTEBROBASILAR INSUFFICIENCY (Nervous system disorders) | 1 (1) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 2 (2) | 0 (0)
URETEROLITHIASIS (Renal and urinary disorders) | 1 (1) | 0 (0)
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 2 (2) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GDC-0853 (200mg BID) Cohort 1 (N=410) | GDC-0853 (200mg BID) Cohort 2 (N=86)
URINARY TRACT INFECTION (Infections and infestations) | 22 (28) | 4 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-08): https://cdn.clinicaltrials.gov/large-docs/27/NCT02983227/Prot_SAP_000.pdf